CLINICAL TRIAL: NCT02616835
Title: Investigating the Physiology of Targeted Theta-burst Neuromodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mental Health Nottingham (Other)
Responsible Party: Principal Investigator, Sarina Iwabuchi, Dr Sarina Iwabuchi, Institute of Mental Health Nottingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: L14082014 SoM PAPsych
Record Dates: First submitted 2015-11-24; First posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- theta-burst TMS (Experimental): Theta-Burst protocol for transcranial magnetic stimulation on dorsolateral prefrontal cortex (exact location to be determined using neuronavigation guided by Magnetic Resonance Imaging)
  Interventions: Device: theta-burst TMS
- sham theta-burst TMS (Sham Comparator): Sham protocol for theta-burst transcranial magnetic stimulation on dorsolateral prefrontal cortex (exact location to be determined using neuronavigation guided by Magnetic Resonance Imaging)
  Interventions: Device: sham theta-burst TMS

INTERVENTIONS:
Device: theta-burst TMS — This protocol involves short periods of pulse delivery in combination with long periods of silent intervals.
  Arms: theta-burst TMS
Device: sham theta-burst TMS — This protocol delivers theta-burst pulses from a sham device (i.e. at same speed and timeframe but without the magnetic output)
  Arms: sham theta-burst TMS

SUMMARY:
This research seeks to study the physiological effects of theta-burst transcranial magnetic stimulation (TMS) in the brains of healthy controls using functional MRI and spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* No personal history of neurological or psychiatric disorders

Exclusion Criteria:

* Have had a brain injury or neurological disorder
* Have ever suffered an epileptic fit
* Have any non-removable metal implants
* Drink more than 20 units of alcohol per week on a regular basis
* Currently take any illicit drugs on regular basis
* Likely to be pregnant
* Ever suffered from a serious mental illness such as schizophrenia, severe depression or bipolar disorder
* Currently take any psychotropic medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Changes in functional connectivity following TMS administration using functional MRI | One hour
  Changes in brain connectivity will be assessed by comparing functional MRI scans after theta-burst TMS and sham theta-burst TMS

SECONDARY OUTCOMES:
Changes in brain metabolites following TMS administration using MR spectroscopy | One hour
  Using MRI scans, changes in metabolites in the brain will be assessed following theta-burst TMS and sham TMS

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Iwabuchi, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Sarina Iwabuchi, Nottingham, Nottinghamshire, United Kingdom